CLINICAL TRIAL: NCT03506334
Title: Prospective Pilot Study of Anterior Vertebral Body Tethering Using Zimmer Biomet Tether System or Dynesys System Components to Treat Pediatric Scoliosis
Brief Title: Anterior Vertebral Body Tethering (AVBT) Using Zimmer Biomet Tether System or Dynesys System Components to Treat Pediatric Scoliosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, MD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-007801
Record Dates: First submitted 2018-04-03; First posted 2018-04-24 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Tether group 40 patients and Fusion (control) group 40 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pediatric Scoliosis Patients (Experimental): Tether group
  Interventions: Device: AVBT using Dynesys System Components
- Pediatric Scoliosis Control Patients (Active Comparator): Fusion (control) group
  Interventions: Procedure: Spine fusion

INTERVENTIONS:
Device: AVBT using Dynesys System Components — Zimmer Biomet Tether System and Dynesys System components are intended to treat scoliosis in skeletally immature children.
  Arms: Pediatric Scoliosis Patients
Procedure: Spine fusion — Children with scoliosis undergoing fusion surgery will form the control arm
  Arms: Pediatric Scoliosis Control Patients

SUMMARY:
The Researchers want to assess the short-term safety of Anterior Vertebral Body Tethering (AVBT) in skeletally immature subjects with moderate to severe scoliosis and compare them with a fusion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male & female, age 10 years to 16 years.
2. Scoliosis curve between 40-70 degrees.
3. At least 1 year of growth remaining measured by Sanders bone age 4 or less or Risser stage 2 or less.
4. Adolescent idiopathic scoliosis.
5. Lenke 1, 2, 3C, 5 (thoracic, thoracolumbar, or thoracic and lumbar).
6. Parents must be able to understand the study and sign the consent document. Assent will be obtained and documented as age appropriate.
7. Patients and parents must be able to comply with study procedures and visits, including 3-month, 1-year, and 2-year follow-up visits.

Exclusion Criteria:

1. Congenital, neuromuscular or syndromic scoliosis.
2. Underlying neuromuscular disease.
3. Pregnancy.
4. Nonflexible curves (bending films show residual curve greater than 40 degrees).
5. Prior surgery for scoliosis treatment.
6. Patients with active systemic infection.
7. Known, reported allergies to titanium, PET, or PCU. Known, reported substance abuse, including alcohol.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Revision spine surgery within 2 years of index procedure | 2 years
  yes/no parameter, was revision surgery performed within 2 years of index procedure

SECONDARY OUTCOMES:
Major cobb angle curve progression greater than 10 degrees and curve magnitude < 50 degrees at latest f/u after 1st erect postop film (Tether arm) | 1 year
  yes/no parameter, did major Cobb angle worsen by 10 degrees and curve magnitude < 50 degrees at latest f/u after 1st erect postop film
Curve progression no greater than 10 degrees at latest f/u after 1st erect postop film (Fusion arm) | 1 year
  yes/no parameter, did major Cobb angle worsen by 10 degrees at latest f/u after 1st erect postop film
Curve flexibility over instrumented vertebra > 5 degrees | At least 1 year postoperatively
  Flexibility films will be obtained in patients postoperatively to assess flexibility
Spinal disc health utilizing MRI | At least 1 year postoperatively
  Spinal disc health will be assessed in Tether patients post-operatively using an MRI in conjunction with the Pfirrmann classification (scored I to V, where I indicated normal and V indicated the worst degeneration).

CONTACTS AND LOCATIONS:
Overall Officials: A. Noelle Larson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathew SE, Hargiss JB, Milbrandt TA, Stans AA, Shaughnessy WJ, Larson AN. Vertebral body tethering compared to posterior spinal fusion for skeletally immature adolescent idiopathic scoliosis patients: preliminary results from a matched case-control study. Spine Deform. 2022 Sep;10(5):1123-1131. doi: 10.1007/s43390-022-00519-3. Epub 2022 May 24. PMID 35610543